CLINICAL TRIAL: NCT06310889
Title: Evaluation of Palliative Care Co-treatment by Attending Physicians and Nurses: an Online Survey as Part of the Project (EPIC-Baseline-Survey)
Brief Title: Evaluation of Palliative Care Co-treatment by Attending Physicians and Nurses: an Online Survey as Part of the Project
Acronym: EPIC-BS
Status: Withdrawn | Type: Observational
Why Stopped: Already registered
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: European Commission (Other); National and Kapodistrian University of Athens (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: EPIC-Baseline-Survey
Record Dates: First submitted 2024-02-22; First posted 2024-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Palliative Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The subject of the study is an online survey of doctors and nurses who provide (intensive) medical care to patients.

DETAILED DESCRIPTION:
Charité will support this international survey as part of the preparatory phase of the "Europe-wide harmonized and recommended palliative care practice for ICU" approved HORIZON grant application EPIC (EA2/291/23), to which this ethics application refers.

Participants will be contacted via the mailing list of ESAIC (European Organization for Anaesthesia, Intensive Care, Pain and Perioperative Medicine), ESICM (European Society of Intensive Care Medicine), DIVI (German Interdisciplinary Association for Intensive Care and Emergency Medicine (DIVI) and the European Association for Palliative Care (EAPC).

ELIGIBILITY:
Inclusion Criteria:

* All doctors or nursing staff involved in the intensive medical care of patients and consent to the survey via the distribution list of a specialist association

Exclusion Criteria:

* Incomplete data

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Doctors or nursing staff involved in the intensive medical care of patients which can be contacted by a list of a specialist association
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Barriers 1 | 01.04.2024 - 30.06.2024
  Barriers in palliative care regarding implementation of therapeutic goals (implementation rate symptom assessment for e.g. breathing and dyspnea).
Barriers 2 | 01.04.2024 - 30.06.2024
  Barriers in palliative care regarding implementation of patient automomy (implementation rate to define advance directives and power of attorney).

SECONDARY OUTCOMES:
Measures 1 | 01.04.2024 - 30.06.2024
  Measures to be taken in the palliative medical treatment situation (implementation rate to define and document end-of-life-decisions).
Measures 2 | 01.04.2024 - 30.06.2024
  Evaluation of measures to be taken in the palliative medical treatment situation (family involvement in end-of-life-decisions).
Resources 1 | 01.04.2024 - 30.06.2024
  Personnel resources in palliative care (rate of specialized palliative care team available in ICUs).
Resources 2 | 01.04.2024 - 30.06.2024
  Other resources in palliative care (rate availability of psychological support)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Chair — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No